CLINICAL TRIAL: NCT05488782
Title: A Pilot RCT of a Remotely Delivered Self-management Program (TEAM-Red) for Depressed Young African American Women at Risk for Hypertension (HTN)
Brief Title: TEAM-Red, a Remotely Delivered Self-management Program for Depressed Black Women at Risk for Hypertension
Acronym: TEAM-Red
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer B. Levin (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor-Investigator, Jennifer B. Levin, Principal Investiagator, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY20220976
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: 41 participants are assigned to receive TEAM, and 41 participants are assigned to wait list
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TEAM-Red (Experimental): Five 60-minute group sessions with 6-10 patients. These sessions will be held weekly and delivered remotely via videoconference
  Interventions: Behavioral: TEAM-Red
- Enhanced Waitlist (eWL) (Other): After the week 12 follow up visit, subjects in the Waitlist group will receive the TEAM Red intervention
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: TEAM-Red — Five 60-minute group sessions with 6-10 patients. These sessions will be held weekly and delivered remotely via videoconference
  Arms: TEAM-Red
Other: Waitlist — After the week 12 follow up visits subjects in the Waitlist group will receive the TEAM Red intervention
  Arms: Enhanced Waitlist (eWL)

SUMMARY:
The proposed project is a 24-week prospective randomized controlled trial (RCT) evaluating the effects of TargEted MAnageMent Intervention (TEAM, N=41) vs. enhanced waitlist (eWL, N=41) control in young (<50 years) African American women who are depressed or suffering from stress, and at risk for hypertension.

ELIGIBILITY:
Phase 1 Inclusion Criteria:

1. Registered on Research Goes Red;
2. Self-identified African American female ages 18-49;
3. current depression as measured by a score of ≥10 on the 9-item Patient Health Questionnaire (PHQ-9),
4. Have at least one of the following self or chart-recorded HTN risk factors: body mass index (BMI) greater ≥ 30, HbA1c >5.75, at least one outpatient reading of systolic blood pressure (BP) ≥ 130 mm Hg or diastolic ≥90 mmHg, current smoker, or LDL ≥100 mg/dl in the last 12 months;
5. Are able to participate in study procedures.

Phase 1 Exclusion Criteria:

1. Unwilling/unable to provide informed consent;
2. Pregnancy;
3. Imminent suicide risk,
4. A current diagnosis of hypertension or use of antihypertensive medications.

Phase 2 Inclusion Criteria

1. Self-identified AA female ages 18-49;
2. Endorses either: a past or current history of depression, current depression as measured by a score of at least a 5 on the 9-item Patient Health Questionnaire (PHQ-9), or indicate feelings of stress or discrimination that impact their functioning
3. Have at least one of the following self or chart-recorded HTN risk factors: BMI greater ≥ 30,26 HbA1c >5.75,27 at least one outpatient reading of systolic BP ≥ 130 mm Hg or diastolic ≥90 mmHg, current smoker, or LDL ≥100 mg/dl in the last 12 months;
4. Are able to participate in study procedures.

Phase 2 Exclusion Criteria

1. Unwilling/unable to provide informed consent;
2. Pregnancy;
3. Imminent suicide risk,
4. A current diagnosis of HTN or use of antihypertensive medications.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 82 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase 1 TEAM vs WL change in 9-item Patient Health Questionnaire (PHQ-9) total score at 12-week follow-up | Baseline to 12 weeks
  PHQ-9 total score ranges from 0 to 27, with a higher score indicating a higher level depression
Phase 1 change in 9-item Patient Health Questionnaire (PHQ-9) total score at 24-week follow up | Baseline to 24 weeks
  PHQ-9 total score ranges from 0 to 27, with a higher score indicating a higher level depression
Phase 2 TEAM-Red vs eWL 9-item Patient Health Questionnaire (PHQ-9) total score at 12-week follow-up | Baseline to 12 weeks
  PHQ-9 total score ranges from 0 to 27, with a higher score indicating a higher level depression
Phase 2 change in 9-item Patient Health Questionnaire (PHQ-9) total score at 24-week follow-up | Baseline to 24 weeks
  PHQ-9 total score ranges from 0 to 27, with a higher score indicating a higher level depression
Phase 2 TEAM-Red vs eWL 10-item Perceived Stress Scale (PSS-10) total score at 12-week follow-up | Baseline to 12 weeks
  PSS-10 total scores ranges from 0 to 40 with a higher score indicating a higher level of perceived stress
Phase 2 change in 10-item Perceived Stress Scale (PSS-10) total score at 24-week follow up | Baseline to 24 weeks
  PSS-10 total scores ranges from 0 to 40 with a higher score indicating a higher level of perceived stress

SECONDARY OUTCOMES:
Phase 1 TEAM-Red vs eWL 10-item Perceived Stress Scale (PSS-10) total score at 12-week follow-up | Baseline to 12 weeks
  PSS-10 total scores ranges from 0 to 40 with a higher score indicating a higher level of perceived stress
Phase 1 change in 10-item Perceived Stress Scale (PSS-10) total score at 24-week follow up | Baseline to 24 weeks
  PSS-10 total scores ranges from 0 to 40 with a higher score indicating a higher level of perceived stress
Phase 1 TEAM-Red vs eWL 12-item Short Form Survey (SF-12) mental component score at 12-week follow up | Baseline to 12 weeks
  SF-12 mental component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to mental health
Phase 1 TEAM-Red vs eWL 12-item Short Form Survey (SF-12) physical component score at 12-week follow up | Baseline to 12 weeks
  SF-12 physical component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to physical health
Phase 1 change in 12-item Short Form Survey (SF-12) mental component score at 24-week follow up | Baseline to 24 weeks
  SF-12 mental component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to mental health
Phase 1 change in 12-item Short Form Survey (SF-12) physical component score at 24-week follow up | Baseline to 24 weeks
  SF-12 physical component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to physical health
Phase 2 TEAM-Red vs eWL change in 12-item Short Form Survey (SF-12) mental component score at 12-week follow-up | Baseline to 12 weeks
  SF-12 mental component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to mental health
Phase 2 TEAM-Red vs eWL change in 12-item Short Form Survey (SF-12) physical component score at 12-week follow-up | Baseline to 12 weeks
  SF-12 physical component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to physical health
Phase 2 change in 12-item Short Form Survey (SF-12) mental component score at 24-week follow up | Baseline to 24 weeks
  SF-12 mental component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to mental health
Phase 2 change in 12-item Short Form Survey (SF-12) physical component score at 24-week follow up | Baseline to 24 weeks
  SF-12 physical component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to physical health
Phase 1 and Phase 2 TEAM-Red vs eWL change in 9-item Patient Health Questionnaire (PHQ-9) total score at 12-week follow-up | Baseline to 12 weeks
  PHQ-9 total score ranges from 0 to 27, with a higher score indicating a higher level depression
Phase 1 and Phase 2 change in 9-item Patient Health Questionnaire (PHQ-9) total score at 24-week follow up | Baseline to 24 weeks
  PHQ-9 total score ranges from 0 to 27, with a higher score indicating a higher level depression
Phase 1 and Phase 2 TEAM-Red vs eWL change in 10-item Perceived Stress Scale (PSS-10) total score at 12-week follow-up | Baseline to 12 weeks
  PSS-10 total scores ranges from 0 to 40 with a higher score indicating a higher level of perceived stress
Phase 1 and Phase 2 change in 10-item Perceived Stress Scale (PSS-10) total score at 24-week follow up | Baseline to 24 weeks
  PSS-10 total scores ranges from 0 to 40 with a higher score indicating a higher level of perceived stress
Phase 1 and Phase 2 TEAM-Red vs eWL change in 12-item Short Form Survey (SF-12) mental component score at 12-week follow-up | Baseline to 12 weeks
  SF-12 mental component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to mental health
Phase 1 and Phase 2 TEAM-Red vs eWL change in 12-item Short Form Survey (SF-12) physical component score at 12-week follow-up | Baseline to 12 weeks
  SF-12 physical component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to physical health
Phase 1 and Phase 2 change in 12-item Short Form Survey (SF-12) mental component score at 24-week follow up | Baseline to 24 weeks
  SF-12 mental component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to mental health
Phase 1 and Phase 2 change in 12-item Short Form Survey (SF-12) physical component score at 24-week follow up | Baseline to 24 weeks
  SF-12 physical component score ranges from 0 to 100, with higher scores indicating a better quality of life as it relates to physical health

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Levin, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data with the data dictionary and protocol will be made available to other researchers via the American Heart Association (AHA) Precision Medicine Platform
Supporting Information: Study Protocol
Time Frame: Data will be available by one year following the funding